CLINICAL TRIAL: NCT02712528
Title: Recovery Profiles of Remifentanil-based vs. Sevoflurane-sufentanil Combined Regimen for Cardiac Surgery
Brief Title: Recovery Profiles of Remifentanil-based Regimen for Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH1160080
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Cardiac Surgery
Keywords: bispectral index; extubation; recovery; remifentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil-based (Active Comparator): remifentanil-based regimen consisting of remifentanil 0.75 mcg/kg/min and supplemental propofol for maintaining BIS 40-60
  Interventions: Drug: remifentanil-based
- sevoflurane-sufentanil balanced (Placebo Comparator): balanced sevoflurane (end-tidal 1.2-2.8 vol%) and sufentanil (0.015 mcg/kg/min) regimen
  Interventions: Drug: sevoflurane-sufentanil balanced

INTERVENTIONS:
Drug: remifentanil-based
  Arms: remifentanil-based
Drug: sevoflurane-sufentanil balanced
  Arms: sevoflurane-sufentanil balanced

SUMMARY:
Backgrounds: Monitoring of Bispectral index (BIS) has been regarded as useful to determine the degree of intraoperative hypnosis. Major factors of postoperative recovery after cardiac surgery include patient's recovery in cognitive function from the postoperative residual effects of anesthetics, such as opioids and sedatives, administered during intraoperative period. Therefore employing anesthetic regimens which can provide earlier recovery in cognitive function would be beneficial in facilitating fast-track cardiac surgery with earlier postoperative extubation and discharge from the intensive care unit (ICU).

Previous investigations suggested efficacy of BIS in evaluating the degree of postoperative hypnosis in the ICU.

The present study compares the time for reaching BIS greater than 80 after using 2 different anesthesia regimens for cardiac surgery, remifentanil-based regimen and sevoflurane-sufentanil balanced regimen.

Analyzing the changes immediately after cardiac surgery would be useful to determine the degree of patient's postoperative emergence.

Materials and Methods:

During study period, patients undergoing elective cardiac surgery in Konkuk University Medical Center are randomly assigned to get remifentanil-based regimen consisting of remifentanil 0.75 mcg/kg/min and supplemental propofol for maintaining BIS 40-60 (Group R) or sevoflurane (end-tidal 1.2-2.8 vol%) and sufentanil (0.015 mcg/kg/min) balanced regimen in Group S.

All patients get intravenous patient controlled anesthesia consisting of alfentanyl and ondansetron after surgery. Supplemental remifentanil 0.25-0.3 mcg/kg/min is administered during postoperative 2 hours in Group R.

As a primary objective, inter-group difference in the time for achieving BIS greater than 80 is determined.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective coronary artery bypass surgery

Exclusion Criteria:

* combined valve surgery
* preoperative intraaortic balloon pumping
* preoperative low cardiac output syndrome
* chronic obstructive pulmonary disease

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to reach BIS > 80 | 1 minute
  Time to reach BIS > 80 after surgery

SECONDARY OUTCOMES:
Extubation time | 1 minute
  Time to perform extubation after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yop Kim, MD, PhD, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No